CLINICAL TRIAL: NCT05619484
Title: Smart Ankle-Foot Orthosis to Improve Stroke Outcomes: Smart AFO
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Orthocare Innovations, LLC (Industry)
Collaborators: Becker Orthopedic (Unknown); University of Utah (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 0019-01
Record Dates: First submitted 2022-10-10; First posted 2022-11-17 (Actual); Last update posted 2023-10-10 (Actual); Status verified 2023-10

CONDITIONS: Stroke
Keywords: ankle-foot orthosis; orthotist
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Participant's prescribed ankle-foot orthosis (No Intervention)
- Smart AFO (Experimental)
  Interventions: Device: Smart AFO

INTERVENTIONS:
Device: Smart AFO — Diagnostic ankle-foot orthosis with AFO stiffness and range of motion settings adjusted using a mobile application
  Arms: Smart AFO

SUMMARY:
The Smart Ankle-Foot Orthosis (Smart AFO) system is an investigational system that combines a diagnostic ankle-foot orthosis with a mobile application to assist clinicians in optimizing an AFO user's gait by adjusting AFO stiffness and range of motion settings, and quantifying functional walking improvements in post-stroke individuals. The purpose of the clinical testing is to evaluate the Smart AFO system with its target users: post-stroke AFO users and orthotists. This may include, but is not limited to, identifying any aspects of the Smart AFO system that could be improved through clinical testing and evaluating the gait of post-stroke AFO users walking with an AFO adjusted using the Smart AFO system.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Mass less than 90 kg (200 lbs)
* At least six months post-stroke
* Hemiplegia or hemiparesis as a result of stroke
* Foot drop during swing phase (often identified by a toe catch), on at least one side
* Current user of an AFO
* Current user of an AFO with a Triple Action Joint is acceptable
* Has bilateral passive ankle range of motion within normal limits
* Able to walk safely on level ground for at least 100 feet without rest
* Able to communicate individual perceptions in the English language
* Able to provide written informed consent
* Participants that will use a treadmill during data collection must also be able to walk independently and safely on an instrumented treadmill

Exclusion Criteria:

* Confounding injury, musculoskeletal issues, or cognitive issues that limit effective participation
* Pregnancy
* Not able to read and understand English
* Use of assistive device that requires bilateral upper extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-08-15 (Actual); Primary Completion 2024-08-31 (Estimated); Study Completion 2024-08-31 (Estimated)

PRIMARY OUTCOMES:
Timed Up and Go (TUG) test | Assessed on day 1 (data collection day) with prescribed AFO
  The Timed Up and Go (TUG) test is a validated timed functional test that involves standing up from a chair, walking forward for 3 meters, turning around, walking back to the chair for 3 meter, and sitting down. Measured in seconds.
Timed Up and Go (TUG) test | Assessed on day 1 (data collection day) with Smart AFO
  The Timed Up and Go (TUG) test is a validated timed functional test that involves standing up from a chair, walking forward for 3 meters, turning around, walking back to the chair for 3 meter, and sitting down. Measured in seconds.
Ankle plantarflexion | Assessed on day 1 (data collection day) with prescribed AFO
  Average ankle joint angle at foot flat after initial contact (degrees)
Ankle plantarflexion | Assessed on day 1 (data collection day) with Smart AFO
  Average ankle joint angle at foot flat after initial contact (degrees)
Ankle power | Assessed on day 1 (data collection day) with prescribed AFO
  Average peak ankle joint power during stance phase (Newton-meters/second)
Ankle power | Assessed on day 1 (data collection day) with Smart AFO
  Average peak ankle joint power during stance phase (Newton-meters/second)
Knee angle | Assessed on day 1 (data collection day) with prescribed AFO
  Average knee joint angle at midstance (degrees)
Knee angle | Assessed on day 1 (data collection day) with Smart AFO
  Average knee joint angle at midstance (degrees)
Knee power | Assessed on day 1 (data collection day) with prescribed AFO
  Average knee joint power at foot flat after initial contact (Newton-meters/second)
Knee power | Assessed on day 1 (data collection day) with Smart AFO
  Average knee joint power at foot flat after initial contact (Newton-meters/second)
Ankle dorsiflexion | Assessed on day 1 (data collection day) with prescribed AFO
  Average ankle joint angle during midswing (degrees)
Ankle dorsiflexion | Assessed on day 1 (data collection day) with Smart AFO
  Average ankle joint angle during midswing (degrees)

SECONDARY OUTCOMES:
Stride length | Assessed on day 1 (data collection day) with prescribed AFO
  Average stride length of steps (meters)
Stride length | Assessed on day 1 (data collection day) with Smart AFO
  Average stride length of steps (meters)

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Becker Orthopedic, Troy, Michigan
  - University of Utah, Salt Lake City, Utah
  - Orthocare Innovations, LLC, Edmonds, Washington

IPD SHARING:
Plan to Share IPD: No